CLINICAL TRIAL: NCT06386393
Title: Survey on Where Parents Look for and Find Information and How They Use Information When Selecting Child Care
Status: Completed | Type: Observational
Sponsor: National Opinion Research Center (Other)
Collaborators: Office of Planning, Research & Evaluation (U.S. Federal Agency); Urban Institute (Other)
Responsible Party: Principal Investigator, Rupa Datta, Vice President and Distinguished Senior Fellow, National Opinion Research Center
Other Study IDs: HHSP233201500048I-75P00120F370
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Searching for and Selecting Child Care in the US
Keywords: consumer education strategies; child care and early education search; surveys

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Administration for Children and Families (ACF) within the U.S. Department of Health and Human Services (HHS) is contracting with NORC at the University of Chicago to collect nationally representative survey data to learn more about where parents look for and find information about Child Care and Early Education (CCEE); how parents assess the people, places, or things that may offer CCEE information; what types of CCEE information parents look for; and how parents use information to make CCEE selections. The study aims to gather information that may be used by Child Care Lead Agencies to inform their consumer education efforts. This study is part of the Consumer Education and Parental Choice in Early Care and Education (CEPC) project.

The study will select a nationally representative sample from NORC's probability-based AmeriSpeak panel. The AmeriSpeak panel provides sample coverage of approximately 97 percent of the U.S. population. It currently contains 48,900 panel members age 13 and over residing in over 40,000 households. U.S. households are randomly selected with a known, non-zero probability from the NORC National Frame, and then recruited by mail, telephone, and by field interviewers face-to-face. NORC's in-person recruitment enhances representativeness for young adults, lower socio-economic households, non-internet households, and other households that are typically hard to reach for statistical surveys of the population.

The survey respondents are AmeriSpeak panelists of at least 18 years of age who have indicated that they have a young child in the household (under the age of 6 years, but not in kindergarten). If a household has two or more panel members who reside in a household with a young child, one will be selected at random to complete the survey, with preference given to parents/legal guardians. Selected panelists will be asked questions to confirm eligibility for the survey, including that the household has at least one child under the age of 6 but not in kindergarten. The study is designed to include parents and legal guardians across race/ethnicity, education level, and gender from the full spectrum of geographic locations. To include families who may not have English as a preferred language, a Spanish version of the survey will be provided. The survey will include parents and legal guardians using many kinds of CCEE and those who use parental care only to see if there are differences in how information is used depending on care type. In addition, the study will include understudied subgroups, such as parents who speak a language other than English, to help inform consumer education efforts. The survey is intended to produce findings that are generalizable to the larger population of parents with children under the age of 6, but not in kindergarten.

DETAILED DESCRIPTION:
Aims: The primary purpose of the study is to collect nationally representative survey data to learn more about where parents look for and find information about Child Care and Early Education (CCEE); how parents assess the people, places, or things that may offer CCEE information; what types of CCEE information parents look for; and how parents use information to select CCEE. The study aims to gather information that may be used by Child Care Lead Agencies to inform their consumer education efforts.

The project will select a nationally representative sample from NORC's probability-based AmeriSpeak panel. The AmeriSpeak panel provides sample coverage of approximately 97 percent of the U.S. population. It currently contains 48,900 panel members age 13 and over residing in over 40,000 households. U.S. households are randomly selected with a known, non-zero probability from the NORC National Frame, and then recruited by mail, telephone, and by field interviewers face-to-face. NORC's in-person recruitment enhances representativeness for young adults, lower socio-economic households, non-internet households, and other households that are typically hard to reach for statistical surveys of the population.

The survey will collect information about (a) where parents look for and find information about CCEE; (b) how parents assess the people, places, or things that may offer CCEE information; (c) how easy or hard it is for parents to find CCEE information, (d) the types of CCEE information that parents look for and say are helpful in choosing CCEE; (e) information about the last time parents made a decision about CCEE and what information they tried to learn about at that time; (f) parent's assessments of the CCEE options at the time they made their last CCEE decision; (g) how well parents' CCEE decision met their family's needs; and (h) demographic information about families. The survey is intended to produce findings that are generalizable to the larger population of parents with children under the age of 6, but not in kindergarten. This survey will provide insights on how child care lead agencies can reach parents searching for CCEE and to share consumer education information.

The study will address the following research questions:

1. Where do parents search for and find information about CCEE options (e.g., family, friends, states' and territories' consumer education)?
2. What types of information are parents searching for before making decisions about CCEE for their children?
3. How do parents evaluate the information they find or come across about possible CCEE options?
4. How do parents use the information they find or come across to inform the decisions they make about CCEE?
5. What characteristics of CCEE programs are most salient to their decision-making process?
6. What are key facilitators and barriers to parents' finding and/or using consumer information?

Recruitment and data collection. Participants: Respondents for this study will include AmeriSpeak panelists who indicated that they have a young child in the household. Panelists will be invited to complete the survey if they are at least 18 years of age. If a household has two or more panel members who reside in a household with a young child, only one panelist will be selected at random to complete the survey, with preference given to parents/legal guardians. Selected panelists will be asked questions to confirm eligibility for the survey, including that the household has at least one child under the age of 6 but not in kindergarten. Data will be collected beginning in March 2024. The investigators will recruit panelists using multiple contact modes (email, mail, phone, and SMS text messages where appropriate). Data will be collected through an online web survey or by an AmeriSpeak interviewer over the phone. Both will be available in English and Spanish.

Data Analysis. The analytic focus of the study is to document and identify patterns in parents' knowledge and use of different sources of information during their CCEE search and selection process. The investigators will also document and explore parent perspectives and experiences with using different information sources on CCEE, including the challenges parents face when they try to find information about CCEE. The investigators will begin analysis by creating key variables of interest (individual survey items and/or factors) and inspecting their distributions and rates of missingness. If contextual information from other data sources is required (e.g., about local characteristics or information about state consumer-education resources), the investigators will prepare those variables during data collection to have available for analysis. For example, the investigators may use American Community Survey (ACS) or similar external data sources to better understand the communities where households live. Because the main analytic objective is descriptive in nature, statistics will be focused on weighted frequencies, means, and proportions.

ELIGIBILITY:
Inclusion Criteria:

* Survey of AmeriSpeak panelists of at least 18 years of age who have indicated that they have a young child in the household (under the age of 6 years, but not in kindergarten).
* If a household has two or more panel members who reside in a household with a young child, one will be selected at random to complete the survey, with preference given to parents/legal guardians.
* Selected panelists will be asked questions to confirm eligibility for the survey, including that the household has at least one child under the age of 6 but not in kindergarten.

Exclusion Criteria:

• Being under the age of 18 and not having children under the age of 6 years that are not in kindergarten

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AmeriSpeak panelists who indicated that they have a young child in the household and who are at least 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 6804 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Primary sources of information about child care | March-June 2024
  The parent survey will collect information about where parents may have gotten information from or tried to get information about CCEE.
How parents assess the people, places, or things that may offer CCEE information | March-June 2024
  The parent survey will collect information about how parents rate different sources of information including whether the source is current, has specific information they want to know, makes it easy to find information, and is trustworthy.
What types of CCEE related information parents look for | March-June 2024
  The parent survey will collect information on what child care and early education information parents have looked for within the last twelve months, what information they found most helpful, and information they have not found but think would be most helpful about child care options in their area.
Information about the last time parents made a decision about CCEE and what information they tried to learn about at that time | March-June 2024
  The parent survey will collect information about the main reason parents made their last CCEE decision, how many hours they spent looking for information to help make a decision, how many weeks they had to consider information before making a CCEE decision, whether they considered one or more providers when making a decision, the specific information they tried to learn when they made that decision, whether parents think they had enough information when they made that decision, whether the families had no options or had one or more options for child care, how well the decision met their family's needs, and whether as a result of the decision if they had to make changes to their work or family situation.

SECONDARY OUTCOMES:
Characteristics and experiences of the household and types of CCEE being used | March-June 2024
  The parent survey will also collect information about the household, including demographic information (i.e., the state the parent or guardian lives in, household income, work schedules) and about the types of CCEE care being used including use of non-parental care, paid or unpaid center-based or home-based care.

CONTACTS AND LOCATIONS:
Overall Officials: Rupa Datta, PhD, Principal Investigator — NORC at the University of Chicago
Locations (1):
- NORC at the University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No